CLINICAL TRIAL: NCT03127982
Title: Effects of the Adaptation of the Unified Protocol for Emotional Problems in Victims of the Armed Conflict in Colombia: A Randomized Clinical Trial
Brief Title: Unified Protocol for Emotional Problems in Victims of the Armed Conflict in Colombia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Los Andes, Columbia (Other)
Responsible Party: Principal Investigator, Leonidas Castro Camacho, Ph.D.,ABPP, Associate Professor, University of Los Andes, Columbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: COLCIENCIAS 644-2014
Record Dates: First submitted 2017-04-07; First posted 2017-04-25 (Actual); Last update posted 2022-11-18 (Actual); Status verified 2022-11

CONDITIONS: Emotional Disorder
Keywords: Anxiety Depression Emotion PTSD Randomized Clinical Trial

STUDY DESIGN:
Intervention Model Description: Allocation: Randomized Intervention Model: Parallel Assignment Single Blind
Who Masked: Care Provider, Outcomes Assessor
Masking Description: The clinical staff participating in the intervention are unaware of the group membership of the subjects; either experimental or wait-list.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Immediately following randomization, participants in this condition attend 12-13 biweekly face-to face individual sessions that last approximately 1.5 hrs each of the cultural adaptation of the Unified Protocol trans diagnostic treatment comprising the following modules: motivation enhancement, psycho-education of emotion, emotion awareness training, cognitive reappraisal, emotion avoidance and emotion-driven behavior, tolerance training for physical sensations, emotion exposure, and relapse prevention. Treatment is provided by graduate students in clinical psychology who have been trained in the UP and receive weekly supervision by experienced clinicians and use a Workbook for homework assigned between sessions.
  Interventions: Behavioral: Unified Protocol
- Group 2 (Active Comparator): Participants randomly assigned to this condition do not receive any active intervention during a six-week wait period after randomization, while completing assessment evaluation at the beginning and end of wait list period, after which they receive the same intervention (Unified Protocol) provided to the treatment condition (Group 1).
  Interventions: Behavioral: Unified Protocol

INTERVENTIONS:
Behavioral: Unified Protocol — The Unified Protocol (UP) is a trans-diagnostic cognitive-behavioral therapy (tCBT) for individuals diagnosed with anxiety disorders, depression and related disorders (which we refer to as emotional disorders).
  Other Names: UP for the Transdiagnostic Treatment of Emotional Disorders

SUMMARY:
The present study aims at evaluating the effects of a CBT intervention, a cultural adaptation of the Unified Protocol for the Trans-diagnostic Treatment of Emotional Disorders (UP) in victims of the Colombian armed conflict.

A randomized clinical trial aimed at evaluating the effects of the UP in a group of 100 internally displaced victims of armed conflict living in Bogotá is being implemented. Participants are recruited from several governmental, non-governmental agencies as well as community organizations of victims. Participants are being randomly assigned to treatment condition (N=50) or to waiting-list control (N=50). Treatment consists in 12 biweekly sessions covering the 8 modules of the original UP. The effects of the UP is evaluated through Patient Health Questionnaire (PHQ) and several measures of co-morbid emotional disorders, Anxiety, Depression, PTSD as well as level of functioning and quality of life.

DETAILED DESCRIPTION:
Specific objectives

* To translate and adapt the UP, taking into account the cultural, social, economic and political context of individuals exposed to political violence in Colombia.
* Develop and adapt a set of assessment tools to identify victim's symptoms of anxiety, depression, and related disorders.
* Conduct a randomized clinical trial comparing outcomes of 12 biweekly sessions of the culturally adapted UP in a group participants randomized to immediate treatment to a waiting list control receiving delayed (6-week) treatment.
* To identify potential variables that mediate or moderate the effects of treatment with the UP.

Methodology Design. Allocation randomized Participants. 100 individuals presenting emotional sequelae of exposure to violent events of armed conflict in Colombia, 50 of which are being randomly assigned to treatment group and 50 to control group (waiting list).

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria. Individuals registered as victims in Colombian Victims Unit, 18 years or older, who meet the diagnostic criteria for one or more anxiety disorder(s), depressive disorder(s) or post-traumatic stress and related disorder(s) according to the Diagnostic and Statistical Manual (DSM-5, 2013) as determined by the International Neuro-Psychiatric Interview M.I.N.I.

Exclusion Criteria:

* Exclusion criteria. Individuals diagnosed with psychotic disorders, bipolar affective disorders, intellectual disability, dementia, substance abuse (as primary diagnoses, with hospitalization requirement for treatment) as well as individuals who endorse acute suicidal risk. Those that do not meet the inclusion criteria, but are in need of mental health attention, will be referred to entities of the Health System, so that they receive the pertinent treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Based on self-representation.
Enrollment: 109 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2020-12-20 (Actual); Study Completion 2021-12-20 (Actual)

PRIMARY OUTCOMES:
Changes in diagnostic criteria for depression, anxiety, as assessed by the Patient Health Questionnaire. | Administered at baseline, post-treatment - on average 8 weeks after the beginning of treatment, and a 3-month follow-up.
  PHQ - complete.
Change in symptoms of post-traumatic stress as measured by the Post-Traumatic Stress Disorder (PTSD) | Administered at baseline, post-treatment - on average 8 weeks after the beginning of treatment, and a 3-month follow-up.
  Checklist for the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) (PCL-5).

SECONDARY OUTCOMES:
Quality of Life. Self-reported measure assessing the physical health, subjective feelings, leisure activities, social relationships, general activities, satisfaction with medications and life satisfaction. | Administered at baseline, post-treatment - on average 8 weeks after the beginning of treatment, and a 3-month follow-up.
  Quality of Life Enjoyment Questionnaire, Q-LES-Q.
Anxiety measure. | Administered at baseline, post-treatment - on average 8 weeks after the beginning of treatment, and a 3-month follow-up.
  Overall Anxiety Severity and Impairment Scale (OASIS)
Depression measure. | Administered at baseline, post-treatment - on average 8 weeks after the beginning of treatment, and a 3-month follow-up.
  Overall Depression Severity and Impairment Scale. (ODSIS).
Current level of functioning. | Baseline, and 3-month follow-up.
  Current level of functioning measure. Adapted from ACOPLE. (Santaella-Tenorio J, Bonilla- Escobar FJ, Fandiño-Losada A, Bass J, Gutiérrez-Martínez MI, Bolton P. Validating an Instrument for victims of violence in Colombia: Evaluation of Two Community-based Mental Health Interventions for Violence-Displaced Afro-Descendants in Colombia. [Unpublished manuscript]. Colombia: University of Valle, Instituto CISALVA; 2013). -[Time Frame: Baseline, and 3-month follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Leonidas Castro-Camacho, Ph.D., Principal Investigator — Universidad de Los Andes
Locations (1):
- Laboratorio de Psicología Clínica Uniandes - Universidad de Los Andes, Bogotá, DC, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Castro-Camacho L, Barlow DH, Garcia N, Farchione TJ, Idrobo F, Rattner M, Quant DM, Gonzalez L, Moreno JD. Effects of a Contextual Adaptation of the Unified Protocol in Multiple Emotional Disorders in Individuals Exposed to Armed Conflict in Colombia: A Randomized Clinical Trial. JAMA Psychiatry. 2023 Oct 1;80(10):991-999. doi: 10.1001/jamapsychiatry.2023.2392. PMID 37466983